CLINICAL TRIAL: NCT01009892
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalency Study of Codeine Sulfate Tablets Under Fasting and Fed Conditions
Brief Title: Food Effect Study of Codeine Sulfate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CODE-T60-PVFS/FD-1
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — O(6)-codeine methyl ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Codeine Sulfate, 30 mg (Active Comparator): tablet
  Interventions: Drug: Codeine Sulfate
- Codeine Sulfate, 60 mg (Active Comparator): tablet
  Interventions: Drug: Codeine Sulfate
- Codeine Sulfate, 15 mg (Active Comparator): tablet
  Interventions: Drug: Codeine Sulfate

INTERVENTIONS:
Drug: Codeine Sulfate — Tablet

SUMMARY:
The study was designed to assess the effect of food on the absorption of codeine from Roxane Laboratories' 60 mg Codeine Sulfate tablet

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to Codeine Sulfate or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick Bieberdorf, Principal Investigator — CEDRA Clinical Research
Locations (1):
- CEDRA Clinical Research, San Antonio, Texas, United States